CLINICAL TRIAL: NCT02129088
Title: An Open-Label, Single-Dose Study to Assess the Pharmacokinetics, Safety, and Tolerability of Intranasally Administered Esketamine in Healthy Elderly and Adult Subjects
Brief Title: A Pharmacokinetic, Safety and Tolerability Study of Esketamine in Healthy Elderly and Adult Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Janssen Research & Development, LLC (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CR103806; ESKETINTRD1003 (Other: Janssen Research and Development, LLC); 2013-005372-18 (EudraCT Number)
Record Dates: First submitted 2014-04-30; First posted 2014-05-02 (Estimated); Last update posted 2014-07-25 (Estimated); Status verified 2014-07

CONDITIONS: Healthy
Keywords: Healthy; Esketamine; Phase 1; Placebo; Elderly; Adult
MeSH Terms: interventions — Esketamine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Cohort 1 (Experimental): Participants will receive esketamine 14 milligram (mg) as intranasal spray into each nostril on Day 1.
  Interventions: Drug: Esketamine
- Cohort 2 (Experimental): All participants will receive esketamine 14 mg as intranasal spray into each nostril on Day 1 of Period 1 as Treatment A and esketamine 14 mg as intranasal spray followed by intranasal administration of placebo solution after 5 and 10 minutes of esketamine administration into each nostril on Day 1 of Period 2 as Treatment B in a fixed sequence.
  Interventions: Drug: Esketamine; Drug: Placebo

INTERVENTIONS:
Drug: Esketamine — Esketamine 14 mg will be self-administered by participants as intranasal spray into each nostril on Day 1 to cohort 1 and cohort 2 in a fixed sequence.
Drug: Placebo — Placebo will be self-administered as intranasal spray by participants after 5 and 10 minutes of esketamine administration into each nostril on Day 1 of Treatment period 2 to Cohort 2.
  Arms: Cohort 2

SUMMARY:
The purpose of this study is to compare the pharmacokinetics (explores what the body does to the drug), safety and tolerability of esketamine, administered intranasally (administered through the nose) in healthy elderly (Cohort 1) and healthy adult (Cohort 2) participants.

DETAILED DESCRIPTION:
This is a Phase 1, open-label (all people know the identity of the intervention), single-center, and single-dose study of esketamine, in healthy elderly (Cohort 1) and adult (Cohort 2) participants. Cohort 1 will comprise of 14 healthy elderly participants (greater than or equal to [>=] 65 years) with at least 3 participants above >=75 years of age and Cohort 2 will comprise of 20 healthy adult participants (18 to 55 years of age, inclusive). The study comprises of 3 phases: a Screening phase, an open-label Treatment phase (consisting of 1 treatment period for Cohort 1 and 2 treatment periods for Cohort 2), and a Safety follow-up phase. The duration of Screening phase is of 3 weeks; duration of treatment period for cohort 1 is of 3 days and for cohort 2 is 3 - 5 days (In Treatment period 1: 5 days for the first 7 participants who will complete the additional urine and fecal collection up to 72 hours post dose and 3 days for the last 13 participants who will be discharged after 24 hours; in Treatment period 2: 3 days for all participants). A washout period of 5 to 10 days will separate each intranasal esketamine treatment regimen for Cohort 2. All participants in Cohort 1 will receive Treatment A (that is, esketamine 14 milligram [mg] will be self-administered as intranasal spray into each nostril under the direct supervision of the investigator or designee), whereas, all participants in Cohort 2 will receive Treatment A followed by Treatment B (that is, esketamine 14 mg will be self-administered as intranasal spray followed by self-administration of placebo solution after 5 and 10 minutes of esketamine administration into each nostril, under the direct supervision of the investigator or designee) in a fixed sequence. The total esketamine dose will be 28 mg for each regimen. Blood samples will be collected for evaluation of pharmacokinetic parameters pre-dose and until 24 hours post-dose for evaluation of pharmacokinetic parameters. Participants' safety will be monitored throughout the study.

ELIGIBILITY:
Inclusion Criteria:

* Female participant must be postmenopausal (no spontaneous menses for at least 2 years), surgically sterile, abstinent (abstinence is an acceptable means of birth control only if it is already established as the participant's usual and preferred lifestyle), or, if sexually active, be practicing an effective method of birth control (for example, prescription oral contraceptives, contraceptive injections, intrauterine device, double-barrier method, contraceptive patch, male partner sterilization) before entry and throughout the study
* Body mass index (BMI) between 18 and 30 kilogram per square meter (kg/m^2) (inclusive), and body weight not less than 50 kilogram (kg)
* Systolic blood pressure (after the participant is supine for 5 minutes) between 90 and 150 millimeter of mercury (mmHg) (inclusive) and diastolic blood pressure not more than 90 mmHg
* Comfortable with self-administration of intranasal medication and able to follow instructions provided
* A 12-lead electrocardiogram (ECG) consistent with normal cardiac conduction and function

Exclusion Criteria:

* Current significant psychiatric (mental disorders) disorder including but not limited to psychotic (a person exhibiting mental illness), bipolar, major depressive or anxiety disorder
* Clinically significant medical illness including (but not limited to) cardiac arrhythmias (irregular heart beat) or other cardiac disease, hematologic disease, coagulation disorders (including any abnormal bleeding or blood dyscrasias [disorder of blood]), lipid abnormalities, significant pulmonary (having to do with the lungs) disease, including bronchospastic respiratory disease, diabetes mellitus (disorder in which there is decreased insulin in the body or the body's insulin is not effective, resulting in high blood sugar, increased thirst and urine, and many other side effects), renal or hepatic insufficiency, thyroid disease, neurologic disease, infection, hypertension or vascular disorders, kidney or urinary tract disturbances, sleep apnea (breathing problems while sleeping), myasthenia gravis (disorder that causes muscles to get tired quickly), or any other illness that the Investigator considers should exclude the participant or that could interfere with the interpretation of the study results
* Use of any prescription or nonprescription medication, within 14 days before the first scheduled dose of the study drug
* Anatomical or medical conditions that may delay delivery or absorption of study medication (for example. undergone facial reconstructions, structural or functional abnormalities of the nose or upper airway; obstructions or mucosal lesions (any visible local abnormality of the tissues of the skin) of the nostrils or nasal passages; undergone sinus (a depression or cavity formed by a bending or curving) surgery in the previous 2 years; or signs and symptoms of upper respiratory infection, rhinitis, active allergies, or has a history of frequent sinus infections or complications)
* Has an abnormal or deviated nasal septum (when the inner wall separating the two sides of the nose is off to one side) with any 1 or more of the following symptoms: blockage of 1 or both nostrils, nasal congestion (especially 1-sided), frequent nosebleeds, frequent sinus infections, noisy breathing during sleep, facial pain, headaches, and postnasal drip

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 34 (Actual)
Dates: Start 2014-03; Primary Completion 2014-05 (Actual); Study Completion 2014-05 (Actual)

PRIMARY OUTCOMES:
Maximum Plasma Concentration (Cmax) of Esketamine | 0 (pre-dose), 7, 12, 22, 32, 40, 50 minutes; 1, 1.25, 1.5, 2, 3, 4, 6, 9, 12, 18 and 24 hours after study drug administration
  The Cmax is the maximum plasma concentration.
Time to Reach Maximum Concentration (tmax) | 0 (pre-dose), 7, 12, 22, 32, 40, 50 minutes; 1, 1.25, 1.5, 2, 3, 4, 6, 9, 12, 18 and 24 hours after study drug administration
  The tmax is time to reach the maximum observed plasma concentration.
Area Under the Plasma Concentration-Time Curve From Time Zero to Last Quantifiable Time (AUC [0-last]) | 0 (pre-dose), 7, 12, 22, 32, 40, 50 minutes; 1, 1.25, 1.5, 2, 3, 4, 6, 9, 12, 18 and 24 hours after study drug administration
  The AUC (0-last) is the area under the plasma concentration-time curve from time zero to last quantifiable time.
Area Under the Plasma Concentration-Time Curve From Time Zero to Infinite Time (AUC [0-infinity]) | 0 (pre-dose), 7, 12, 22, 32, 40, 50 minutes; 1, 1.25, 1.5, 2, 3, 4, 6, 9, 12, 18 and 24 hours after study drug administration
  The AUC (0-infinity) is the area under the plasma concentration-time curve from time zero to infinite time, calculated as the sum of AUC(0-last) and C(0-last)/lambda(z), wherein AUC(0-last) is area under the plasma concentration-time curve from time zero to last quantifiable time; C(0-last) is the last observed quantifiable concentration; and lambda(z) is elimination rate constant.
Percentage Area Under the Plasma Concentration Curve From Time Zero to Infinite Time (%AUC [0-infinity]) | 0 (pre-dose), 7, 12, 22, 32, 40, 50 minutes; 1, 1.25, 1.5, 2, 3, 4, 6, 9, 12, 18 and 24 hours after study drug administration
  Percentage AUC[0-infinity] is obtained by extrapolation of the concentration-time curve. It is calculated by AUC[0-infinity] minus AUC[0-last] divided by AUC[0-infinity] multiplied by 100.
Elimination Half-Life (t [1/2] Lambda) | 0 (pre-dose), 7, 12, 22, 32, 40, 50 minutes; 1, 1.25, 1.5, 2, 3, 4, 6, 9, 12, 18 and 24 hours after study drug administration
  Elimination half-life (t [1/2] Lambda) is associated with the terminal slope (lambda [z]) of the semi logarithmic drug concentration-time curve, calculated as 0.693/lambda(z).
Rate Constant (Lambda[z]) | 0 (pre-dose), 7, 12, 22, 32, 40, 50 minutes; 1, 1.25, 1.5, 2, 3, 4, 6, 9, 12, 18 and 24 hour after study drug administration
  Lambda(z) is first-order rate constant associated with the terminal portion of the curve, determined as the negative slope of the terminal log-linear phase of the drug concentration-time curve .

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Research & Development, LLC Clinical Trial, Study Director — Janssen Research & Development, LLC
Locations (1):
- Merksem, Belgium

REFERENCES:
- [Derived] Perez-Ruixo C, Rossenu S, Zannikos P, Nandy P, Singh J, Drevets WC, Perez-Ruixo JJ. Population Pharmacokinetics of Esketamine Nasal Spray and its Metabolite Noresketamine in Healthy Subjects and Patients with Treatment-Resistant Depression. Clin Pharmacokinet. 2021 Apr;60(4):501-516. doi: 10.1007/s40262-020-00953-4. Epub 2020 Oct 31. PMID 33128208